CLINICAL TRIAL: NCT02999178
Title: A Double Blind, Randomized, Placebo-controlled Trial Evaluating the Efficacy and Safety of Nintedanib Over 52 Weeks in Patients With Progressive Fibrosing Interstitial Lung Disease (PF-ILD)
Brief Title: Efficacy and Safety of Nintedanib in Patients With Progressive Fibrosing Interstitial Lung Disease (PF-ILD)
Acronym: INBUILD®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.247; 2015-003360-37 (EudraCT Number)
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nintedanib (Experimental)
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib
  Other Names: OVEF
  Arms: Nintedanib
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of the current study is to investigate the efficacy and safety of nintedanib over 52 weeks in patients with Progressive Fibrosing Interstitial Lung Disease (PF-ILD) defined as patients who present with features of diffuse fibrosing lung disease of >10% extent on high-resolution computed tomography (HRCT) and whose lung function and respiratory symptoms or chest imaging have worsened despite treatment with unapproved medications used in clinical practice to treat ILD. There is currently no efficacious treatment available for PF-ILD. Based on its efficacy and safety in Idiopathic Pulmonary Fibrosis (IPF), it is anticipated that Nintedanib will be a new treatment option for patients with PF-ILD.

ELIGIBILITY:
Inclusion criteria:

* Written Informed Consent consistent with International Conference on Harmonisation Harmonised Tripartite Guideline for Good Clinical Practice (ICH-GCP) and local laws signed prior to entry into the study (and prior to any study procedure including shipment of High Resolution Computer Tomography (HRCT) to reviewer).
* Male or female patients aged >= 18 years at Visit 1.
* Patients with physician diagnosed Interstitial Lung Disease (ILD) who fulfil at least one of the following criteria for Progressive Fibrosing Interstitial Lung Disease (PF-ILD) within 24 months of screening visit (Visit 1) despite treatment with unapproved medications used in clinical practice to treat ILD, as assessed by the investigator (refer to Exclusion Criteria):

  * Clinically significant decline in Forced Vital Capacity (FVC) % pred based on a relative decline of >=10%
  * Marginal decline in FVC % pred based on a relative decline of .>=5-<10% combined with worsening of respiratory symptoms
  * Marginal decline in FVC % pred based on a relative decline of >=5-<10% combined with increasing extent of fibrotic changes on chest imaging
  * Worsening of respiratory symptoms as well as increasing extent of fibrotic changes on chest imaging [Note: Changes attributable to comorbidities e.g. infection, heart failure must be excluded. Unapproved medications used in the clinical practice to treat ILD include but are not limited to corticosteroid, azathioprine, mycophenolate mofetil (MMF), n-acetylcysteine (NAC), rituximab, cyclophosphamide, cyclosporine, tacrolimus].
* Fibrosing lung disease on HRCT, defined as reticular abnormality with traction bronchiectasis with or without honeycombing, with disease extent of >10%, performed within 12 months of Visit 1 as confirmed by central readers.
* For patients with underlying Connective Tissue Disease (CTD): stable CTD as defined by no initiation of new therapy or withdrawal of therapy for CTD within 6 weeks prior to Visit 1.
* Carbon Monoxide Diffusion Capacity (DLCO) corrected for Haemoglobin (Hb) [visit 1] ≥ 30% and <80% predicted of normal at Visit 2
* FVC >= 45% predicted at Visit 2

Exclusion criteria:

* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) > 1.5 x Upper Limit of Normal (ULN) at Visit 1
* Bilirubin > 1.5 x ULN at Visit 1
* Creatinine clearance <30 mL/min calculated by Cockcroft-Gault formula at Visit 1 [Note: Laboratory parameters from Visit 1 have to satisfy the laboratory threshold values as shown above. Visit 2 laboratory results will be available only after randomization. In case at Visit 2 the results do no longer satisfy the entry criteria, the Investigator has to decide whether it is justified that the patient remains on study drug. The justification for decision needs to be documented. Laboratory parameters that are found to be abnormal at Visit 1 are allowed to be re-tested (once) if it is thought to be a measurement error (i.e. there was no abnormal result of this test in the recent history of the patient and there is no related clinical sign) or the result of a temporary and reversible medical condition, once that condition is resolved].
* Patients with underlying chronic liver disease (Child Pugh A, B or C hepatic impairment).
* Previous treatment with nintedanib or pirfenidone.
* Other investigational therapy received within 1 month or 6 half-lives (whichever was greater) prior to screening visit (Visit 1).
* Use of any of the following medications for the treatment of Interstitial Lung Disease (ILD): azathioprine (AZA), cyclosporine, MMF, tacrolimus, oral corticosteroids (OCS) >20mg/day and the combination of OCS+AZA+NAC within 4 weeks of Visit 2, cyclophosphamide within 8 weeks of Visit 2, rituximab within 6 months of Visit 2.

Note: Patients whose Rheumatoid Arthritis (RA)/Connective Tissue Disease (CTD) is managed by these medications should not be considered for participation in the current study unless change in RA/CTD medication is medically indicated (see Inclusion Criteria)

* Diagnosis of Idiopathic Pulmonary Fibrosis (IPF) based on American Thoracic Society (ATS)/ European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) 2011 Guidelines.
* Significant Pulmonary Arterial Hypertension (PAH) defined by any of the following:

  * Previous clinical or echocardiographic evidence of significant right heart failure
  * History of right heart catheterization showing a cardiac index <= 2 l/min/m²
  * PAH requiring parenteral therapy with epoprostenol/treprostinil
  * Primary obstructive airway physiology (pre-bronchodilator FEV1/FVC < 0.7 at Visit 1).
  * In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
* Major extrapulmonary physiological restriction (e.g. chest wall abnormality, large pleural effusion)
* Cardiovascular diseases, any of the following:

  * Severe hypertension, uncontrolled under treatment (≥160/100 mmHg), within 6 month of Visit 1
  * Myocardial infarction within 6 months of Visit 1
  * Unstable cardiac angina within 6 months of Visit 1
* Bleeding risk, any of the following:

  * Known genetic predisposition to bleeding.
  * Patients who require

    * Fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, direct thrombin inhibitors, heparin, hirudin)
    * High dose antiplatelet therapy. [Note: Prophylactic low dose heparin or heparin flush as needed for maintenance of an indwelling intravenous device (e.g. enoxaparin 4000 I.U. s.c. per day), as well as prophylactic use of antiplatelet therapy (e.g. acetyl salicylic acid up to 325 mg/day, or clopidogrel at 75 mg/day, or equivalent doses of other antiplatelet therapy) are not prohibited].
  * History of haemorrhagic central nervous system (CNS) event within 12 months of Visit 1.
  * Any of the following within 3 months of Visit 1:

    * Haemoptysis or haematuria
    * Active gastro-intestinal (GI) bleeding or GI - ulcers
    * Major injury or surgery (Investigators judgment).
  * Coagulation parameters: International normalized ratio (INR) >2, prolongation of prothrombin time (PT) and activated partial thromboplastin time (aPTT) by >1.5 x ULN at Visit 1.
* History of thrombotic event (including stroke and transient ischemic attack) within 12 months of Visit 1.
* Known hypersensitivity to the trial medication or its components (i.e. soya lecithin)
* Patients with peanut allergy.
* Other disease that may interfere with testing procedures or in the judgment of the Investigator may interfere with trial participation or may put the patient at risk when participating in this trial.
* Life expectancy for disease other than ILD < 2.5 years (Investigator assessment).
* Planned major surgical procedures.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Women of childbearing potential* not willing or able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly as well as one barrier method for 28 days prior to and 3 months after nintedanib administration. A list of contraception methods meeting these criteria is provided in the patient information.
* In the opinion of the Investigator, active alcohol or drug abuse.
* Patients not able to understand or follow trial procedures including completion of self-administered questionnaires without help. *A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (152):
- United States (51):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Pulmonary and Sleep Specialists, Danbury, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Pulmonary and Sleep of Tampa Bay, Brandon, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Pulmonary and Critical Care Associates of Baltimore, Towson, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Pulmonary and Critical Care Medicine, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Creighton University, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Oaks, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Pul & Crit Care Conslt, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Medical Arts and Research Center (MARC), San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
- Argentina (6):
  - Centro Dr. Lazaro Langer S.R.L, Alberdi Sur
  - Centro de Investigaciones Metabólicas (CINME), C.a.b.a
  - Sanatorio Güemes, Ciudad Autónoma de Bs As
  - CEMER-Centro Medico De Enfermedades Respiratorias, Florida
  - INSARES, Mendoza
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
- Belgium (4):
  - Centre Hospitalier Universitaire de Liège, Angleur
  - ULB Hopital Erasme, Brussels
  - UZ Leuven, Leuven
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Canada (4):
  - Concordia Hospital, Winnipeg, Manitoba
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CHUS Fleurimont, Sherbrooke, Quebec
- Chile (3):
  - Hospital Clínico Reg. de Concepción "Dr. G. Grant Benavente", Concepción
  - Instituto Nacional del Tórax, Providencia, Santiago de Chile
  - Centro de Investigación del Maule, Talca
- China (4):
  - Peking Union Medical College Hospital, Beijing
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Hospital of Chinese Medical University, Shenyang
- France (13):
  - HOP Avicenne, Bobigny
  - HOP Louis Pradel, Bron
  - HOP Côte de Nacre, Caen
  - HOP d'Instruction des Armées Percy, Clamart
  - HOP Calmette, Lille
  - HOP Nord, Marseille
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Pasteur, Nice
  - HOP Bichat, Paris
  - HOP Maison Blanche, Reims
  - HOP Pontchaillou, Rennes
  - HOP Civil, Strasbourg
  - HOP Bretonneau, Tours
- Germany (9):
  - Universitätsklinikum Bonn AöR, Bonn
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Klinik Donaustauf, Donaustauf
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Wissenschaftliches Institut Bethanien, Solingen
  - Universitätsklinikum Tübingen, Tübingen
  - Petrus-Krankenhaus, Wuppertal
- Italy (6):
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - Ospedale "G.B. Morgagni - L. Pierantoni" ausl forli, Forlì
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - A.O. San Gerardo di Monza, Monza
  - Policlinico Gemelli, Roma
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (20):
  - Tosei General Hospital, Aichi, Seto
  - Kurume University Hospital, Fukuoka, Kurume
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - National Hospital Organization Himeji Medical Center, Hyogo, Himeji
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - Ibarakihigashi National Hospial, Ibaraki, Naka-gun
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Miyagi, Sendai
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Osaka Medical College Hospital, Osaka, Takatsuki
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Tokushima University Hospital, Tokushima, Tokushima
  - Tokyo Medical and Dental University, Tokyo, Bunkyo-ku
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Toranomon Hospital, Tokyo, Minato-ku
  - JR Tokyo General Hospital, Tokyo, Shibuya-ku
  - Global Health and Medicine Ctr, Tokyo, Shinjuku-ku
- Poland (5):
  - University Clinical Center, Gdansk, Gdansk
  - Leszek Giec Upper-Silesian Med.Cent.Silesian Med.Univ., Katowice
  - Norbert Barlicki University Clinical Hospital No.1, Lodz, Lodz
  - Nat.Instit.of Tuberculosis&LungDiseases,Outpat.Clin,warszawa, Warsaw
  - Clinical Hospital No. 1, n.a. Prof. Szyszko from Silesian MA, Zabrze
- Russia (6):
  - Res.Inst.-Compl.Iss.Cardi.Dis., Kemerovo
  - Pulmonology Scientific Research Institute, Moscow
  - Central Scientific Research Insitute of Tuberculosis, Moscow
  - Moscow 1st State Med.Univ.n.a.I.M.Sechenov, Moscow
  - Scientific Research Institute of Pulmonology, Saint Petersburg
  - Emergency Clinical Hospital n. a. N. V. Solovyev, Yaroslavl, Yaroslavl
- South Korea (3):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
- Spain (12):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital de Galdakao, Galdakao
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital La Princesa, Madrid
  - Hospital La Paz, Madrid
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Hospital de Canarias, San Cristóbal de La Laguna
  - Hospital Virgen del Rocío, Seville
  - Hospital Politècnic La Fe, Valencia
- United Kingdom (6):
  - University Hospital Llandough, Cardiff
  - Royal Infirmary of Edinburgh, Edinburgh
  - St James's University Hospital, Leeds
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Royal Stoke University Hospital, Stoke-on-Trent

REFERENCES:
- [Derived] Kolb M, Flaherty KR, Silva RS, Prasse A, Vancheri C, Mueller H, Sroka-Saidi K, Wells AU; INBUILD trial investigators. Effect of Nintedanib in Patients with Progressive Pulmonary Fibrosis in Subgroups with Differing Baseline Characteristics. Adv Ther. 2023 Dec;40(12):5536-5546. doi: 10.1007/s12325-023-02668-x. Epub 2023 Sep 26. PMID 37751022
- [Derived] Kreuter M, Bendstrup E, Jouneau S, Maher TM, Inoue Y, Miede C, Lievens D, Crestani B. Weight loss and outcomes in subjects with progressive pulmonary fibrosis: data from the INBUILD trial. Respir Res. 2023 Mar 9;24(1):71. doi: 10.1186/s12931-023-02371-z. PMID 36894966
- [Derived] Inoue Y, Wells AU, Song JW, Xu Z, Kitamura H, Suda T, Okamoto M, Muller H, Coeck C, Rohr KB, Kolb M, Brown KK. Nintedanib in Asian patients with progressive fibrosing interstitial lung diseases: Results from the INBUILD trial. Respirology. 2023 May;28(5):465-474. doi: 10.1111/resp.14452. Epub 2023 Jan 15. PMID 36642509
- [Derived] Ogura T, Suda T, Inase N, Nishioka Y, Azuma A, Okamoto M, Takizawa A, Ito T, Rohr KB, Inoue Y. Effects of nintedanib on disease progression and safety in Japanese patients with progressive fibrosing interstitial lung diseases: Further subset analysis from the whole INBUILD trial. Respir Investig. 2022 Nov;60(6):787-797. doi: 10.1016/j.resinv.2022.06.009. Epub 2022 Aug 1. PMID 35927208
- [Derived] Cottin V, Martinez FJ, Jenkins RG, Belperio JA, Kitamura H, Molina-Molina M, Tschoepe I, Coeck C, Lievens D, Costabel U. Safety and tolerability of nintedanib in patients with progressive fibrosing interstitial lung diseases: data from the randomized controlled INBUILD trial. Respir Res. 2022 Apr 7;23(1):85. doi: 10.1186/s12931-022-01974-2. PMID 35392908
- [Derived] Swigris JJ, Bushnell DM, Rohr K, Mueller H, Baldwin M, Inoue Y. Responsiveness and meaningful change thresholds of the Living with Pulmonary Fibrosis (L-PF) questionnaire Dyspnoea and Cough scores in patients with progressive fibrosing interstitial lung diseases. BMJ Open Respir Res. 2022 Mar;9(1):e001167. doi: 10.1136/bmjresp-2021-001167. PMID 35241434
- [Derived] Inoue Y, Suda T, Kitamura H, Okamoto M, Azuma A, Inase N, Kuwana M, Makino S, Nishioka Y, Ogura T, Takizawa A, Ugai H, Stowasser S, Schlenker-Herceg R, Takeuchi T. Efficacy and safety of nintedanib in Japanese patients with progressive fibrosing interstitial lung diseases: Subgroup analysis of the randomised, double-blind, placebo-controlled, phase 3 INBUILD trial. Respir Med. 2021 Oct;187:106574. doi: 10.1016/j.rmed.2021.106574. Epub 2021 Aug 12. PMID 34564020
- [Derived] Flaherty KR, Wells AU, Cottin V, Devaraj A, Inoue Y, Richeldi L, Walsh SLF, Kolb M, Koschel D, Moua T, Stowasser S, Goeldner RG, Schlenker-Herceg R, Brown KK; INBUILD Trial Investigators. Nintedanib in progressive interstitial lung diseases: data from the whole INBUILD trial. Eur Respir J. 2022 Mar 17;59(3):2004538. doi: 10.1183/13993003.04538-2020. Print 2022 Mar. PMID 34475231
- [Derived] Maher TM, Brown KK, Kreuter M, Devaraj A, Walsh SLF, Lancaster LH, Belloli EA, Padilla M, Behr J, Goeldner RG, Tetzlaff K, Schlenker-Herceg R, Flaherty KR; INBUILD trial investigators. Effects of nintedanib by inclusion criteria for progression of interstitial lung disease. Eur Respir J. 2022 Feb 3;59(2):2004587. doi: 10.1183/13993003.04587-2020. Print 2022 Feb. PMID 34210788
- [Derived] Cottin V, Richeldi L, Rosas I, Otaola M, Song JW, Tomassetti S, Wijsenbeek M, Schmitz M, Coeck C, Stowasser S, Schlenker-Herceg R, Kolb M; INBUILD Trial Investigators. Nintedanib and immunomodulatory therapies in progressive fibrosing interstitial lung diseases. Respir Res. 2021 Mar 16;22(1):84. doi: 10.1186/s12931-021-01668-1. PMID 33726766
- [Derived] Brown KK, Martinez FJ, Walsh SLF, Thannickal VJ, Prasse A, Schlenker-Herceg R, Goeldner RG, Clerisme-Beaty E, Tetzlaff K, Cottin V, Wells AU. The natural history of progressive fibrosing interstitial lung diseases. Eur Respir J. 2020 Jun 25;55(6):2000085. doi: 10.1183/13993003.00085-2020. Print 2020 Jun. PMID 32217654
- [Derived] Wells AU, Flaherty KR, Brown KK, Inoue Y, Devaraj A, Richeldi L, Moua T, Crestani B, Wuyts WA, Stowasser S, Quaresma M, Goeldner RG, Schlenker-Herceg R, Kolb M; INBUILD trial investigators. Nintedanib in patients with progressive fibrosing interstitial lung diseases-subgroup analyses by interstitial lung disease diagnosis in the INBUILD trial: a randomised, double-blind, placebo-controlled, parallel-group trial. Lancet Respir Med. 2020 May;8(5):453-460. doi: 10.1016/S2213-2600(20)30036-9. Epub 2020 Mar 5. PMID 32145830
- [Derived] Flaherty KR, Wells AU, Cottin V, Devaraj A, Walsh SLF, Inoue Y, Richeldi L, Kolb M, Tetzlaff K, Stowasser S, Coeck C, Clerisme-Beaty E, Rosenstock B, Quaresma M, Haeufel T, Goeldner RG, Schlenker-Herceg R, Brown KK; INBUILD Trial Investigators. Nintedanib in Progressive Fibrosing Interstitial Lung Diseases. N Engl J Med. 2019 Oct 31;381(18):1718-1727. doi: 10.1056/NEJMoa1908681. Epub 2019 Sep 29. PMID 31566307
- [Derived] Flaherty KR, Brown KK, Wells AU, Clerisme-Beaty E, Collard HR, Cottin V, Devaraj A, Inoue Y, Le Maulf F, Richeldi L, Schmidt H, Walsh S, Mezzanotte W, Schlenker-Herceg R. Design of the PF-ILD trial: a double-blind, randomised, placebo-controlled phase III trial of nintedanib in patients with progressive fibrosing interstitial lung disease. BMJ Open Respir Res. 2017 Sep 17;4(1):e000212. doi: 10.1136/bmjresp-2017-000212. eCollection 2017. PMID 29018526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized (1:1 ratio), placebo-controlled, double-blind, parallel-group trial comparing nintedanib to placebo over a 52-week treatment period (Part A). Participants continued on blinded, randomized treatment beyond 52 weeks (Part B). Data base lock (DBL) one was on 6-June-2019, DBL two was on 11-September-2019. Overall Study Period=Part A and B.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 150 mg Nintedanib: 150 milligram (mg) Nintedanib as soft gelatine capsule, administered orally, twice daily (bid), with optional dose reduction to 100 mg bid to manage adverse events (AEs). Continuous daily dosing over a 52-week treatment period (Part A). After completion of the 52-week treatment period, participants continued on blinded treatment until the end of the trial or until a reason for treatment withdrawal was met (Part B).
- Placebo: 150 mg Nintedanib matching placebo, soft gelatine capsule, administered orally, bid, with optional dose reduction to 100 mg bid to manage AEs. Continuous daily dosing over a 52-week treatment period (Part A). After completion of the 52-week treatment period, participants continued on blinded treatment until the end of the trial or until a reason for treatment withdrawal was met (Part B).
Period: Overall Study
Arm/Group | 150 mg Nintedanib | Placebo
Started | 332 | 331
Completed | 218 (On treatment at analysis cut-off date, 12-August-2019) | 231 (On treatment at analysis cut-off date, 12-August-2019)
Not Completed | 114 | 100
Not completed — Adverse Event | 85 | 62
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 21 | 21
Not completed — Other reason not defined above | 7 | 13

BASELINE CHARACTERISTICS:
Population: Treated set: This set included all randomized participants who received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg Nintedanib | Placebo | Total
Number analyzed (Participants) | 332 | 331 | 663
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (9.7) | 66.3 (9.8) | 65.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 154 | 307
  Male | 179 | 177 | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 49 | 96
  Not Hispanic or Latino | 285 | 282 | 567
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 83 | 80 | 163
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 5 | 10
  White | 242 | 246 | 488
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Baseline High Resolution Computed Tomography (HRCT) fibrotic pattern [Count of Participants; unit: Participants] — HRCT fibrotic pattern, i.e. imaging pattern of the lung disease on high-resolution computed tomography assessed by central review. HRCT fibrotic pattern had two categories: 'Usual Interstitial Pneumonia (UIP)-like fibrotic pattern only', 'Other fibrotic patterns'.
  Participants
    UIP-like fibrotic pattern only | 206 | 206 | 412
    Other fibrotic patterns | 126 | 125 | 251
Baseline Forced Vital Capacity (FVC) - Overall Population [Mean (Standard Deviation); unit: Milliliter (mL)] — FVC is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible.
  Milliliter (mL) | 2340.07 (740.19) | 2321.15 (727.97) | 2330.62 (733.62)
Baseline FVC - Participants with HRCT fibrotic pattern=UIP-like fibrotic pattern only [Mean (Standard Deviation); unit: Milliliter (mL)] — FVC is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. Population: All randomized participants with HRCT fibrotic pattern=UIP-like fibrotic pattern only who received at least 1 dose of trial medication.
  Milliliter (mL)
    number analyzed (Participants) | 206 | 206 | 412
    (all) | 2363.43 (762.89) | 2373.59 (720.05) | 2368.51 (740.89)

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Decline in Forced Vital Capacity - Overall Population
Description: Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. Overall population consists of all randomized participants with HRCT fibrotic pattern=UIP-like fibrotic pattern only or HRCT fibrotic pattern= Other fibrotic patterns. Annual rate of decline in Forced Vital Capacity in milliliter (mL) per year in the overall population is based on a random coefficient regression with fixed effects for treatment, HRCT fibrotic pattern, and baseline FVC [mL], and including treatment-by-time and baseline-by-time interactions. Within-participant errors are modelled by an unstructured variance-covariance matrix.
Time Frame: Baseline, 2, 4, 6, 12, 24, 36, 52 weeks after first drug intake (planned post-baseline visits)
Population: All randomized participants in the overall population who received at least 1 dose of trial medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliliter per year
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 332 | 331
Milliliter per year | -80.82 [-110.42 to -51.22] | -187.78 [-216.92 to -158.64]
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; The decrease in FVC was assumed to be linear within each participant over 52 weeks. The intercepts and slopes were assumed to be normally distributed with unstructured covariance matrix. The within participant error was assumed to be independent and normally distributed with mean 0 and a common variance. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors (SEs); Test type: Superiority; p < .0001, Mixed Models Analysis — Treatment comparison of slopes was assessed through the treatment-by-time interaction coefficient. P-value was not adjusted for multiple comparisons; Fixed effects: Treatment, HRCT fibrotic pattern, baseline FVC (mL), treatment-by-time, baseline-by-time interactions. Random effects: time, intercept; Adjusted mean difference = 106.96, 95% CI 2-sided [65.42 to 148.50], Standard Error of Mean 21.15 — Difference of adjusted annual rates of decline was calculated as Nintedanib - Placebo

2. Primary Outcome: Annual Rate of Decline in Forced Vital Capacity - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. Annual rate of decline in Forced Vital Capacity in milliliter (mL) per year in participants with HRCT fibrotic pattern=UIP-like fibrotic pattern only is based on a random coefficient regression with fixed effects for treatment, baseline FVC [mL], and including treatment-by-time and baseline-by-time interactions. Within-participant errors are modelled by an unstructured variance-covariance matrix.
Time Frame: Baseline, 2, 4, 6, 12, 24, 36, 52 weeks after first drug intake (planned post-baseline visits)
Population: All randomized participants with HRCT fibrotic pattern=UIP-like fibrotic pattern only who received at least 1 dose of trial medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliliter per year
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 206 | 206
Milliliter per year | -82.87 [-123.73 to -42.02] | -211.07 [-251.38 to -170.77]
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Fixed effects: Treatment, baseline FVC (mL), treatment-by-time, baseline-by-time interactions. Random effects: time, intercept; Adjusted mean difference = 128.20, 95% CI 2-sided [70.81 to 185.59], Standard Error of Mean 29.17 — Difference of adjusted annual rates of decline was calculated as Nintedanib - Placebo

3. Secondary Outcome: Absolute Change From Baseline in King's Brief Interstitial Lung Disease Questionnaire (K-BILD) Total Score at Week 52 - Overall Population
Description: King's Brief Interstitial Lung Disease questionnaire (K-BILD) consists of 15 items and 3 domains: breathlessness and activities, psychological, and chest symptoms. Possible score ranges from 0-100, score of 100 representing the best health status. If missing items were >50% per domain, the domain score was set to missing. If any of the domain scores were missing, the total score was set to missing. Absolute change from baseline in K-BILD Total score at week 52 in the overall population was based on a Mixed Model Repeated Measures (MMRM), with fixed effects for baseline K-BILD Total score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline-by-visit interactions and random effect for participant. Visit was the repeated measure. Within-participant errors were modelled by unstructured variance-covariance matrix.
Time Frame: Baseline, 12, 24, 36, 52 weeks after first drug intake (planned post-baseline visits)
Population: All randomized participants in the overall population who received at least 1 dose of trial medication and contributed to the model evaluation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 332 | 330
Unit on scale | 0.55 [-0.62 to 1.72] | -0.79 [-1.94 to 0.37]
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; p = 0.1115, Mixed Model Repeated Measures (MMRM); Fixed effects: baseline K-BILD Total score, visit, treatment-by-visit and baseline-by-visit interactions, random effect: participant; Adjusted mean difference = 1.34, 95% CI 2-sided [-0.31 to 2.98], Standard Error of Mean 0.84 — Adjusted mean difference was calculated as Nintedanib - Placebo

4. Secondary Outcome: Absolute Change From Baseline in King's Brief Interstitial Lung Disease (K-BILD) Questionnaire Total Score at Week 52 - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: King's Brief Interstitial Lung Disease questionnaire (K-BILD) consists of 15 items and 3 domains: breathlessness and activities, psychological, and chest symptoms. Possible score ranges from 0-100, score of 100 representing the best health status. If missing items were >50% per domain, the domain score was set to missing. If any of the domain scores were missing, the total score was set to missing. Absolute change from baseline in K-BILD Total score at week 52 in participants with HRCT fibrotic pattern=UIP-like fibrotic pattern only was based on a Mixed Model Repeated Measures (MMRM), with fixed effects for baseline K-BILD Total score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline-by-visit interactions and random effect for participant. Visit was the repeated measure. Within-participant errors were modelled by unstructured variance-covariance matrix.
Time Frame: Baseline, 12, 24, 36, 52 weeks after first drug intake (planned post-baseline visits)
Population: All randomized participants with HRCT fibrotic pattern=UIP-like fibrotic pattern only who received at least 1 dose of trial medication and who contributed to the model evaluation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 206 | 205
Unit on scale | 0.75 [-0.82 to 2.31] | -0.78 [-2.34 to 0.78]
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; p = 0.1747, Mixed Model Repeated Measures (MMRM); [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = 1.53, 95% CI 2-sided [-0.68 to 3.74], Standard Error of Mean 1.12 — Adjusted mean difference was calculated as Nintedanib - Placebo

5. Secondary Outcome: Time to First Acute Interstitial Lung Disease (ILD) Exacerbation or Death Over 52 Weeks - Overall Population
Description: Time to first acute ILD exacerbation or death over 52 weeks was defined as time to first acute ILD exacerbation or death due to any cause within the first 52 weeks and was computed as earliest of date of first documented acute ILD exacerbation or death - date of first drug intake + 1. Participants alive who did not experience any ILD exacerbation event or with unknown status within the first 52 weeks were censored.
Time Frame: From first drug intake until date of first acute ILD exacerbation or date of death or last contact date, up to 372 days
Population: All randomized participants in the overall population who received at least 1 dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 332 | 331
Days | NA [NA to NA] — Non-calculable because the 25 percentile was not reached. | NA [NA to NA] — Non-calculable because the 25 percentile was not reached.
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; p = 0.3948, Log Rank; Stratified by HRCT fibrotic pattern; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.48 to 1.34] — A Cox proportional hazards model, stratified by HRCT fibrotic pattern, was used to estimate the hazard ratio calculated as Nintedanib divided by Placebo

6. Secondary Outcome: Time to First Acute Interstitial Lung Disease (ILD) Exacerbation or Death Over 52 Weeks - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: as for outcome 5
Time Frame: From first drug intake until date of first acute ILD exacerbation or date of death or last contact date, up to 372 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 206 | 206
Days | NA [NA to NA] — Non-calculable because the 25 percentile was not reached. | NA [NA to NA] — Non-calculable because the 25 percentile was not reached.
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; p = 0.1985, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.36 to 1.24] — A Cox proportional hazards model was used to estimate the hazard ratio calculated as Nintedanib divided by Placebo

7. Secondary Outcome: Time to Death Over 52 Weeks - Overall Population
Description: Time to death over 52 weeks defined as the time from date of first drug intake until date of death from any cause for participants with known date of death (from any cause) within the first 52 weeks. Participants with no event (death from any cause) or unknown status within the first 52 weeks were censored.
Time Frame: From first drug intake until date of death or last contact date, up to 372 days
Population: All randomized participants in the overall population who received at least 1 dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 332 | 331
Days | NA [NA to NA] — Non-calculable because the 25 percentile was not reached. | NA [NA to NA] — Non-calculable because the 25 percentile was not reached.
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; p = 0.8544, Log Rank; Stratified by HRCT fibrotic pattern; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.47 to 1.86] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Time to Death Over 52 Weeks - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: as for outcome 7
Time Frame: From first drug intake until date of death or last contact date, up to 372 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 206 | 206
Days | NA [NA to NA] — Non-calculable because the 25 percentile was not reached. | NA [NA to NA] — Non-calculable because the 25 percentile was not reached.
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; p = 0.3291, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.32 to 1.47] — A Cox proportional hazards model was used to estimate the hazard ratio calculated as Nintedanib divided by Placebo

9. Secondary Outcome: Time to Death Due to Respiratory Cause Over 52 Weeks - Overall Population
Description: Time to death due to respiratory cause over 52 weeks is defined as the time from date of first drug intake until date of death attributed to respiratory causes (determined by an independent Adjudication Committee) for participants with known date of death (from respiratory causes) within the first 52 weeks. Participants with no event (death from respiratory causes) or unknown status within the first 52 weeks were censored. As less than 4.95% of the total of participants in the analysis population experienced an event, only descriptive statistics were performed, as pre-specified.
Time Frame: From date of first trial drug intake up to date of death from respiratory causes or last contact date, up to 372 days
Population: All randomized participants in the overall population who received at least 1 dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 332 | 331
Days | NA [NA to NA] — Non-calculable because the 25 percentile was not reached. | NA [NA to NA] — Non-calculable because the 25 percentile was not reached.

10. Secondary Outcome: Time to Death Due to Respiratory Cause Over 52 Weeks - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: as for outcome 9
Time Frame: From date of first trial drug intake up to date of death from respiratory causes or last contact date, up to 372 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 206 | 206
Days | NA [NA to NA] — Non-calculable because the 25 percentile was not reached. | NA [NA to NA] — Non-calculable because the 25 percentile was not reached.

11. Secondary Outcome: Time to Progression or Death Over 52 Weeks - Overall Population
Description: Time to progression or death over 52 weeks is defined as the time from date of first drug intake to date of progression, or date of death (from any cause) if a participant died earlier. Participants with no event (progression or death from any cause) or unknown status were censored. Date of progression is defined as the date when ≥ 10% of absolute decline in FVC percent predicted compared to baseline occured for the first time. Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. Predicted normal values of FVC were calculated according to the Global Lung Initiative. FVC percent predicted (FVC % pred) is the FVC divided by its predicted value in percent.
Time Frame: From first drug intake until date of progression or date of death or last contact date, up to 372 days
Population: All randomized participants in the overall population who received at least 1 dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 332 | 331
Days | NA [367 to NA] — Non-calculable because the 50 percentile was not reached. | NA [269 to NA] — Non-calculable because the 50 percentile was not reached.
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; p = 0.0017, Log Rank; Stratified by HRCT fibrotic pattern; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.49 to 0.85] — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Time to Progression or Death Over 52 Weeks - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: as for outcome 11
Time Frame: From first drug intake until date of progression or date of death or last contact date, up to 372 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 206 | 206
Days | NA [365 to NA] — Non-calculable because the 50 percentile was not reached. | NA [254 to NA] — Non-calculable because the 50 percentile was not reached.
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; p = 0.0081, Log Rank; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.45 to 0.89] — A Cox proportional hazards model was used to estimate the hazard ratio calculated as Nintedanib divided by Placebo

13. Secondary Outcome: Percentage of Participants With a Relative Decline From Baseline in FVC Percent Predicted of More Than 10 Percent at Week 52 - Overall Population
Description: Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. Predicted normal values of FVC were calculated according to the Global Lung Initiative. FVC percent predicted (FVC % pred) is the FVC divided by its predicted value in percent. Participants with relative decline from baseline in FVC % pred greater than 10% at week 52 were those participants with a negative relative change from baseline in FVC % pred at week 52 the absolute value of which being greater than 10% and those participants with missing data (worst case analysis).
Time Frame: Baseline and up to 52 weeks after first drug intake
Population: All randomized participants in the overall population who received at least 1 dose of trial medication.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 332 | 331
Percentage of participants | 40.7 | 48.9
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; Regression, Logistic; Logistic regression model with continuous covariate baseline FVC % pred and binary covariate HRCT fibrotic pattern; Adjusted Odds Ratio = 0.70, 95% CI 2-sided [0.52 to 0.96] — Ratio calculated as Nintedanib divided by Placebo

14. Secondary Outcome: Percentage of Participants With a Relative Decline From Baseline in FVC Percent Predicted of More Than 10 Percent at Week 52 - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: as for outcome 13
Time Frame: Baseline and up to 52 weeks after first drug intake
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 206 | 206
Percentage of participants | 41.3 | 52.4
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; Regression, Logistic; Logistic regression model with continuous covariate baseline FVC % pred; Adjusted Odds Ratio = 0.63, 95% CI 2-sided [0.43 to 0.94] — Ratio calculated as Nintedanib divided by Placebo

15. Secondary Outcome: Percentage of Participants With a Relative Decline From Baseline in FVC Percent Predicted of More Than 5 Percent at Week 52 - Overall Population
Description: Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. Predicted normal values of FVC were calculated according to the Global Lung Initiative. FVC percent predicted (FVC % pred) is the FVC divided by its predicted value in percent. Participants with relative decline from baseline in FVC % pred greater than 5% at week 52 were those participants with a negative relative change from baseline in FVC % pred at week 52 the absolute value of which being greater than 5% and those participants with missing data (worst case analysis).
Time Frame: Baseline and up to 52 weeks after first drug intake
Population: All randomized participants in the overall population who received at least 1 dose of trial medication.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 332 | 331
Percentage of participants | 52.4 | 68.6
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; Regression, Logistic; Logistic regression model with continuous covariate baseline FVC % pred and binary covariate HRCT fibrotic pattern; Adjusted Odds Ratio = 0.50, 95% CI 2-sided [0.36 to 0.68] — Ratio calculated as Nintedanib divided by Placebo

16. Secondary Outcome: Percentage of Participants With a Relative Decline From Baseline in FVC Percent Predicted of More Than 5 Percent at Week 52 - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: as for outcome 15
Time Frame: Baseline and up to 52 weeks after first drug intake
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 206 | 206
Percentage of participants | 52.4 | 70.4
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; Regression, Logistic; Logistic regression model with continuous covariate baseline FVC % pred; Adjusted Odds Ratio = 0.46, 95% CI 2-sided [0.31 to 0.69] — Ratio calculated as Nintedanib divided by Placebo

17. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Symptoms Dyspnea Domain Score at Week 52 - Overall Population
Description: Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms dyspnea domain score (dyspnea score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in dyspnea score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline dyspnea score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline dyspnea score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analysed participants in the model (not only participants with a baseline and measurement at week 52).
Time Frame: Baseline, 12, 24, 36, 52 weeks after first drug intake (planned post-baseline visits)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 329 | 323
Unit on scale | 4.28 [2.43 to 6.14] | 7.81 [5.97 to 9.66]
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; Mixed Model Repeated Measures; Fixed effects: baseline, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline-by-visit interaction, random effect: participant; Adjusted mean difference = -3.53, 95% CI 2-sided [-6.14 to -0.92], Standard Error of Mean 1.33 — Adjusted mean difference was calculated as Nintedanib - Placebo

18. Secondary Outcome: Absolute Change From Baseline in L-PF Symptoms Dyspnea Domain Score at Week 52 - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms dyspnea domain score (dyspnea score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in dyspnea score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline dyspnea score, visit, treatment-by-visit interaction, baseline dyspnea score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analysed participants in the model (not only participants with a baseline and measurement at week 52).
Time Frame: Baseline, 12, 24, 36, 52 weeks after first drug intake (planned post-baseline visits)
Population: All randomized participants with HRCT fibrotic pattern=UIP-like fibrotic pattern only who received at least 1 dose of trial medication and contributed to the model evaluation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 204 | 201
Unit on scale | 4.14 [1.81 to 6.47] | 8.32 [5.99 to 10.66]
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; Mixed Model Repeated Measures; Fixed effects: baseline, visit, treatment-by-visit interaction, baseline-by-visit interaction, random effect: participant; Adjusted mean difference = -4.18, 95% CI 2-sided [-7.48 to -0.88], Standard Error of Mean 1.68 — Adjusted mean difference was calculated as Nintedanib - Placebo

19. Secondary Outcome: Absolute Change From Baseline in L-PF Symptoms Cough Domain Score at Week 52 - Overall Population
Description: Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms cough domain score (cough score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in cough score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline cough score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline cough score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analysed participants in the model (not only participants with a baseline and measurement at week 52).
Time Frame: Baseline, 12, 24, 36, 52 weeks after first drug intake (planned post-baseline visits)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 327 | 320
Unit on scale | -1.84 [-4.36 to 0.69] | 4.25 [1.74 to 6.76]
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; Mixed Model Repeated Measures; [statistical method as in outcome 17, analysis 1]; Adjusted mean difference = -6.09, 95% CI 2-sided [-9.65 to -2.53], Standard Error of Mean 1.81 — Adjusted mean difference was calculated as Nintedanib - Placebo

20. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Symptoms Cough Domain Score at Week 52 - Participants With HRCT Fibrotic Pattern=UIP-like Fibrotic Pattern Only
Description: Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms cough domain score (cough score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in cough score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline cough score, visit, treatment-by-visit interaction, baseline cough score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analysed participants in the model (not only participants with a baseline and measurement at week 52).
Time Frame: Baseline, 12, 24, 36, 52 weeks after first drug intake (planned post-baseline visits)
Population: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | 150 mg Nintedanib | Placebo
Number analyzed (Participants) | 203 | 199
Unit on scale | -3.20 [-6.43 to 0.04] | 4.09 [0.85 to 7.32]
Statistical Analysis 1: Comparison: 150 mg Nintedanib vs Placebo; Test type: Other — No formal hypotheses were tested; Mixed Model Repeated Measures; [statistical method as in outcome 18, analysis 1]; Adjusted mean difference = -7.28, 95% CI 2-sided [-11.86 to -2.71], Standard Error of Mean 2.33 — Adjusted mean difference was calculated as Nintedanib - Placebo

ADVERSE EVENTS:
Time Frame: Treatment period plus 28 days (residual effect period), up to 836 days. Time frame for All-Cause-Mortality: Treatment period plus Follow-up, up to 900 days.
Description: All participants who signed the informed consent.
Groups:
- Nintedanib: 150 milligram (mg) Nintedanib as soft gelatine capsule, administered orally, twice daily (bid), with optional dose reduction to 100 mg bid to manage adverse events (AEs). Continuous daily dosing over a 52-week treatment period (Part A). After completion of the 52-week treatment period, participants continued on blinded treatment until the end of the trial or until a reason for treatment withdrawal was met (Part B).
Arm/Group | Nintedanib | Placebo
All-Cause Mortality (participants affected / at risk) | 36/332 | 45/331
Serious Adverse Events (participants affected / at risk) | 147/332 | 164/331
Other Adverse Events (participants affected / at risk) | 308/332 | 266/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=332) | Placebo (N=331)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 3 | 1
Angina pectoris (Cardiac disorders) | 2 | 3
Angina unstable (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 1
Atrial flutter (Cardiac disorders) | 1 | 2
Atrial thrombosis (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 2
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Chronic right ventricular failure (Cardiac disorders) | 0 | 1
Cor pulmonale acute (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 3
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Long QT syndrome (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Systolic anterior motion of mitral valve (Cardiac disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Mixed deafness (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 2
Glaucoma (Eye disorders) | 1 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal vascular thrombosis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Cardiac death (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Condition aggravated (General disorders) | 2 | 1
Death (General disorders) | 1 | 0
Discomfort (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 6 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Liver injury (Hepatobiliary disorders) | 3 | 2
Adenovirus infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 4 | 5
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 2
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Encephalitis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 2
Herpes zoster oticus (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 4 | 4
Leishmaniasis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 3 | 3
Meningitis aseptic (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Pneumococcal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 24 | 16
Pneumonia bacterial (Infections and infestations) | 1 | 3
Pneumonia legionella (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 3
Pneumonia viral (Infections and infestations) | 0 | 2
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 3
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Electrocardiogram Q wave abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 1
Rotavirus test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 2
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Winged scapula (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Hypokinesia (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 3
Anxiety disorder (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Eosinophilic pneumonia chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 19 | 45
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Arteritis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 2
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 2 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=332) | Placebo (N=331)
Abdominal pain (Gastrointestinal disorders) | 34 | 9
Abdominal pain upper (Gastrointestinal disorders) | 33 | 6
Constipation (Gastrointestinal disorders) | 25 | 32
Diarrhoea (Gastrointestinal disorders) | 239 | 85
Nausea (Gastrointestinal disorders) | 100 | 33
Vomiting (Gastrointestinal disorders) | 64 | 16
Asthenia (General disorders) | 18 | 14
Chest pain (General disorders) | 17 | 14
Fatigue (General disorders) | 34 | 21
Oedema peripheral (General disorders) | 18 | 22
Pyrexia (General disorders) | 17 | 18
Hepatic function abnormal (Hepatobiliary disorders) | 19 | 3
Bronchitis (Infections and infestations) | 44 | 62
Nasopharyngitis (Infections and infestations) | 54 | 48
Respiratory tract infection (Infections and infestations) | 18 | 12
Upper respiratory tract infection (Infections and infestations) | 26 | 25
Urinary tract infection (Infections and infestations) | 22 | 20
Alanine aminotransferase increased (Investigations) | 47 | 12
Aspartate aminotransferase increased (Investigations) | 41 | 12
Gamma-glutamyltransferase increased (Investigations) | 22 | 6
Weight decreased (Investigations) | 49 | 18
Decreased appetite (Metabolism and nutrition disorders) | 54 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 26
Dizziness (Nervous system disorders) | 19 | 15
Headache (Nervous system disorders) | 37 | 27
Insomnia (Psychiatric disorders) | 18 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 50
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49 | 46
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between Principal Investigators and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02999178/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT02999178/SAP_001.pdf